CLINICAL TRIAL: NCT03702816
Title: The Relationship Between Neuropsychological Testing and MRI, PET and Blood Biomarkers in Neurodegenerative Disease (COBRE - Project 1): AIM 2
Brief Title: The Relationship Between Neuropsychological Testing and MRI, PET and COBRE - Project 1: AIM 2 (GE-180)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: GE180 has limited Blood - brain barrier permeation, reducing its utility in neuroinflammation. COVID19 created supply chain issues, impacting enrollment.
Sponsor: Aaron Ritter, MD (Other)
Responsible Party: Sponsor-Investigator, Aaron Ritter, MD, Director of Clinical Trials, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 15-888
Record Dates: First submitted 2018-10-01; First posted 2018-10-11 (Actual); Results first posted 2023-05-24 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-04

CONDITIONS: Alzheimer Disease; Parkinson Disease; Inflammation
Keywords: neuroinflammation
MeSH Terms: conditions — Alzheimer Disease; Parkinson Disease; Inflammation; Neuroinflammatory Diseases

STUDY DESIGN:
Intervention Model Description: All participants will receive one Flutriciclamide (18F-GE180) PET scan.
Masking Description: No masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Alzheimer's Disease (Experimental): Alzheimer's Disease
  GE180 PET Scan
  Interventions: Drug: GE180 PET Scan
- Parkinson's Disease (Experimental): Parkinson's Disease
  GE180 PET Scan
  Interventions: Drug: GE180 PET Scan
- Control (Experimental): Control Group
  GE180 PET Scan
  Interventions: Drug: GE180 PET Scan
- Mild Cognitive Impairment (Experimental): Mild Cognitive Impairment
  GE180 PET Scan
  Interventions: Drug: GE180 PET Scan

INTERVENTIONS:
Drug: GE180 PET Scan — GE180 PET Scan
  Other Names: Flutriciclamide (F18-GE180)

SUMMARY:
The complex pathological cascades leading to both Alzheimer's disease (AD) and Parkinson's disease (PD) involve, at various points, inflammation. Since inflammation is a treatable symptom, understanding how and when it impacts the brain, and where specifically in the brain, would offer important guidance in the development of new treatments, sorely needed in both diseases.

Microglia play an important anti-inflammatory role, and produce a substance, mitochondrial translocator protein (TSPO), whose presence can be used as a marker of regional inflammation. GE180 is a newly developed PET ligand which binds to TSPO and hence can be used in imaging studies to analyze regional inflammation in living patients. In prior studies it has shown regional specificity in multiple sclerosis and brain injury. In the current study, the investigators will be using GE180 to analyze regional and global inflammation in the brains of patients with AD and PD at a single time point.

The results of the current study will provide enriched understanding of inflammation in these conditions, and potentially provide preliminary data to inform design of future interventional trials.

DETAILED DESCRIPTION:
This study will involve a cohort that is currently being established at the Cleveland Clinic Lou Ruvo Center for Brain Health. The cohort has been established under the NIH Center of Biomedical Research Excellence (COBRE) grant and involves annual collection of detailed neuropsychological testing and biomarkers (blood and neuroimaging) from all participants annually. Data are filed in a registry (CNTN). Participants include healthy controls, participants with PD (with and without mild cognitive impairment (MCI)) and patients with MCI (with or without positive florbetapir scan, which demonstrates underlying AD changes likely causing the cognitive impairment) and patients with AD. For the current study, we will focus on patients with MCI with associated underlying AD or PD.

Participants will undergo GE180 PET one time during the study. The approach to PET data collection and analysis will be similar to work done previously with an earlier generation ligand (Edison et al., 2008) and to other work with this tracer (Fan et al., 2016). Participants will complete ECGs and have their vitals taken prior to and immediately following injections. Briefly, the ligand will be injected, there will be a 90 minute uptake period, and scan acquisition will commence for 30 minutes, and will be collected in list mode and rebinned into 18 time frames post acquisition.

The total duration of the study visit will be around 4 hours, and the participants will receive $50 compensation for the visit.

ELIGIBILITY:
Inclusion Criteria:

1. Be enrolled in CNTN
2. Aged 55 to 90
3. Available study partners
4. Willing and able to participate in longitudinal follow-up study
5. For MCI patients, fit criteria based in Movement Disorders Task Force or NIA

Exclusion Criteria:

1. Significant neurological disorders other than AD or PD;
2. Unstable medical conditions
3. History of major psychiatric diseases
4. MRI evidence of infarction or other focal lesion or multiple lacunes
5. Clinically significant abnormalities in B12 or TSH
6. Identified as having a common polymorphism (rs6971) in the TSPO gene which has been shown to reduce binding affinity of tracers similar to GE180. This testing will be done as part of their CNTN participation.

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-12-13 (Actual); Primary Completion 2019-09-29 (Actual); Study Completion 2019-09-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aaron R Ritter, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Lou Ruvo Center for Brain Health, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maphis N, Xu G, Kokiko-Cochran ON, Jiang S, Cardona A, Ransohoff RM, Lamb BT, Bhaskar K. Reactive microglia drive tau pathology and contribute to the spreading of pathological tau in the brain. Brain. 2015 Jun;138(Pt 6):1738-55. doi: 10.1093/brain/awv081. Epub 2015 Mar 31. PMID 25833819
- [Background] Kim YS, Joh TH. Microglia, major player in the brain inflammation: their roles in the pathogenesis of Parkinson's disease. Exp Mol Med. 2006 Aug 31;38(4):333-47. doi: 10.1038/emm.2006.40. PMID 16953112
- [Background] Ji K, Miyauchi J, Tsirka SE. Microglia: an active player in the regulation of synaptic activity. Neural Plast. 2013;2013:627325. doi: 10.1155/2013/627325. Epub 2013 Nov 3. PMID 24303218
- [Background] Benavides J, Fage D, Carter C, Scatton B. Peripheral type benzodiazepine binding sites are a sensitive indirect index of neuronal damage. Brain Res. 1987 Sep 22;421(1-2):167-72. doi: 10.1016/0006-8993(87)91287-x. PMID 2891401
- [Background] Fan Z, Calsolaro V, Atkinson RA, Femminella GD, Waldman A, Buckley C, Trigg W, Brooks DJ, Hinz R, Edison P. Flutriciclamide (18F-GE180) PET: First-in-Human PET Study of Novel Third-Generation In Vivo Marker of Human Translocator Protein. J Nucl Med. 2016 Nov;57(11):1753-1759. doi: 10.2967/jnumed.115.169078. Epub 2016 Jun 3. PMID 27261523
- [Background] Chauveau F, Boutin H, Van Camp N, Dolle F, Tavitian B. Nuclear imaging of neuroinflammation: a comprehensive review of [11C]PK11195 challengers. Eur J Nucl Med Mol Imaging. 2008 Dec;35(12):2304-19. doi: 10.1007/s00259-008-0908-9. Epub 2008 Oct 1. PMID 18828015
- [Background] Boutin H, Murray K, Pradillo J, Maroy R, Smigova A, Gerhard A, Jones PA, Trigg W. 18F-GE-180: a novel TSPO radiotracer compared to 11C-R-PK11195 in a preclinical model of stroke. Eur J Nucl Med Mol Imaging. 2015 Mar;42(3):503-11. doi: 10.1007/s00259-014-2939-8. Epub 2014 Oct 29. PMID 25351507
- [Background] Liu B, Le KX, Park MA, Wang S, Belanger AP, Dubey S, Frost JL, Holton P, Reiser V, Jones PA, Trigg W, Di Carli MF, Lemere CA. In Vivo Detection of Age- and Disease-Related Increases in Neuroinflammation by 18F-GE180 TSPO MicroPET Imaging in Wild-Type and Alzheimer's Transgenic Mice. J Neurosci. 2015 Nov 25;35(47):15716-30. doi: 10.1523/JNEUROSCI.0996-15.2015. PMID 26609163
- [Background] Calsolaro V, Edison P. Neuroinflammation in Alzheimer's disease: Current evidence and future directions. Alzheimers Dement. 2016 Jun;12(6):719-32. doi: 10.1016/j.jalz.2016.02.010. Epub 2016 May 11. PMID 27179961
- [Background] Edison P, Archer HA, Gerhard A, Hinz R, Pavese N, Turkheimer FE, Hammers A, Tai YF, Fox N, Kennedy A, Rossor M, Brooks DJ. Microglia, amyloid, and cognition in Alzheimer's disease: An [11C](R)PK11195-PET and [11C]PIB-PET study. Neurobiol Dis. 2008 Dec;32(3):412-9. doi: 10.1016/j.nbd.2008.08.001. Epub 2008 Aug 15. PMID 18786637
- [Background] Owen DR, Yeo AJ, Gunn RN, Song K, Wadsworth G, Lewis A, Rhodes C, Pulford DJ, Bennacef I, Parker CA, StJean PL, Cardon LR, Mooser VE, Matthews PM, Rabiner EA, Rubio JP. An 18-kDa translocator protein (TSPO) polymorphism explains differences in binding affinity of the PET radioligand PBR28. J Cereb Blood Flow Metab. 2012 Jan;32(1):1-5. doi: 10.1038/jcbfm.2011.147. Epub 2011 Oct 19. PMID 22008728
- [Background] Yokokura M, Mori N, Yagi S, Yoshikawa E, Kikuchi M, Yoshihara Y, Wakuda T, Sugihara G, Takebayashi K, Suda S, Iwata Y, Ueki T, Tsuchiya KJ, Suzuki K, Nakamura K, Ouchi Y. In vivo changes in microglial activation and amyloid deposits in brain regions with hypometabolism in Alzheimer's disease. Eur J Nucl Med Mol Imaging. 2011 Feb;38(2):343-51. doi: 10.1007/s00259-010-1612-0. Epub 2010 Sep 16. PMID 20844871
- [Background] Dickens AM, Vainio S, Marjamaki P, Johansson J, Lehtiniemi P, Rokka J, Rinne J, Solin O, Haaparanta-Solin M, Jones PA, Trigg W, Anthony DC, Airas L. Detection of microglial activation in an acute model of neuroinflammation using PET and radiotracers 11C-(R)-PK11195 and 18F-GE-180. J Nucl Med. 2014 Mar;55(3):466-72. doi: 10.2967/jnumed.113.125625. Epub 2014 Feb 10. PMID 24516258
- [Background] Turkheimer FE, Rizzo G, Bloomfield PS, Howes O, Zanotti-Fregonara P, Bertoldo A, Veronese M. The methodology of TSPO imaging with positron emission tomography. Biochem Soc Trans. 2015 Aug;43(4):586-92. doi: 10.1042/BST20150058. Epub 2015 Aug 3. PMID 26551697
- [Background] Rizzo G, Veronese M, Tonietto M, Zanotti-Fregonara P, Turkheimer FE, Bertoldo A. Kinetic modeling without accounting for the vascular component impairs the quantification of [(11)C]PBR28 brain PET data. J Cereb Blood Flow Metab. 2014 Jun;34(6):1060-9. doi: 10.1038/jcbfm.2014.55. Epub 2014 Mar 26. PMID 24667911

RESULTS

PARTICIPANT FLOW:
Groups:
- Control: Control Group
  GE180 PET Scan, 2 μg/mL IV, 185MBq
- Mild Cognitive Impairment: Mild Cognitive Impairment
  GE180 PET Scan, 2 μg/mL IV, 185MBq
- Alzheimer's Disease: Alzheimer's Disease
  GE180 PET Scan, 2 μg/mL IV, 185MBq
- Parkinson's Disease: Parkinson's Disease
  GE180 PET Scan, 2 μg/mL IV, 185MBq
Period: Overall Study
Arm/Group | Control | Mild Cognitive Impairment | Alzheimer's Disease | Parkinson's Disease
Started | 10 | 7 | 3 | 4
Completed | 10 | 7 | 3 | 4
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Mild Cognitive Impairment | Alzheimer's Disease | Parkinson's Disease | Total
Number analyzed (Participants) | 10 | 7 | 3 | 4 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 1 | 1 | 0 | 5
  >=65 years | 7 | 6 | 2 | 4 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.6 (7.96) | 75.7 (11.22) | 74 (10.23) | 74.7 (3.49) | 72.2 (8.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 2 | 0 | 10
  Male | 5 | 4 | 1 | 4 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 9 | 7 | 3 | 4 | 23
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 0 | 1
  White | 7 | 6 | 3 | 4 | 20
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 0 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 10 | 7 | 3 | 4 | 24

OUTCOME MEASURES:

1. Primary Outcome: Frontal GE180 Standardized Uptake Value Ratio (SUVR)
Description: Frontal SUVR- GE180 binding potential in the frontal cortical ROI, as a marker of frontal neuroinflammation. Frontal neuroinflammation would be expected to relate to frontal lobe AD pathology, and given known frontal lobe role in executive system function, is hypothesized to relate to measures of executive function in particular, and also to memory and language dysfunction, as these have executive components. Greater frontal lobe GE180 is expected to relate to poorer cognitive function.
Time Frame: Baseline (Single scan)
Measure: Mean (Standard Deviation); unit: SUVR
Arm/Group | Control | Mild Cognitive Impairment | Alzheimer's Disease | Parkinson's Disease
Number analyzed (Participants) | 10 | 7 | 3 | 4
SUVR | 0.8893 (0.058) | 0.9436 (0.055) | 0.8855 (0.036) | 0.8850 (0.049)
Statistical Analysis 1: Comparison: Control; Linear Regression of Memory Composite Scores and Frontal GE180 SUVR in Control Subjects; Test type: Other — Linear Regression; p = 0.60, Regression, Linear; F=0.308
Statistical Analysis 2: Comparison: Control; Linear Regression of Executive Function Composite Scores and Frontal GE180 SUVR in Control Subjects; Test type: Other — Linear Regression; p = 0.56, Regression, Linear; F=0.367
Statistical Analysis 3: Comparison: Control; Linear Regression of Speed Composite Scores and Frontal GE180 SUVR in Control Subjects; Test type: Other — Linear regression; p = 0.44, Regression, Linear
Statistical Analysis 4: Comparison: Control; Linear Regression of Language Composite Scores and Frontal GE180 SUVR in Control Subjects; Test type: Other — Linear Regression; p = 0.15, Regression, Linear; F=2.55
Statistical Analysis 5: Comparison: Mild Cognitive Impairment; Linear Regression of Memory Composite Scores and Frontal GE180 SUVR in MCI Subjects; Test type: Other — Linear Regression; p = 0.39, Regression, Linear; F=0.947
Statistical Analysis 6: Comparison: Mild Cognitive Impairment; Linear Regression of Executive Function Composite Scores and Frontal GE180 SUVR in MCI Subjects; Test type: Other — Linear Regression; p = 0.95, Regression, Linear; F=0.004
Statistical Analysis 7: Comparison: Mild Cognitive Impairment; Linear Regression of Speed Composite Scores and Frontal GE180 SUVR in MCI Subjects; Test type: Other — Linear Regulation; p = 0.53, Regression, Linear; F=0.483
Statistical Analysis 8: Comparison: Mild Cognitive Impairment; Linear Regression of Language Composite Scores and Frontal GE180 SUVR in MCI Subjects; Test type: Other — Linear Regression; p = 0.19, Regression, Linear; F=2.543
Statistical Analysis 9: Comparison: Alzheimer's Disease; Linear Regression of Memory Composite Scores and Frontal GE180 SUVR in AD Subjects; Test type: Other — Linear Regression; p = 0.32, Regression, Linear; F=3.430
Statistical Analysis 10: Comparison: Alzheimer's Disease; Linear Regression of Executive Function Composite Scores and Frontal GE180 SUVR in AD Subjects; Test type: Other — Linear Regression; p = 0.11, Regression, Linear; F=32.844
Statistical Analysis 11: Comparison: Alzheimer's Disease; Linear Regression of Speed Composite Scores and Frontal GE180 SUVR in AD Subjects; Test type: Other — Linear Regression; p = 0.31, Regression, Linear; F=3.559
Statistical Analysis 12: Comparison: Alzheimer's Disease; Linear Regression of Language Composite Scores and Frontal GE180 SUVR in AD Subjects; Test type: Other — Linear Regression; p = 0.005, Regression, Linear; F=14362.699
Statistical Analysis 13: Comparison: Parkinson's Disease; Linear Regression of Memory Composite Scores and Frontal GE180 SUVR in PD Subjects; Test type: Other — Linear Regression; p = 0.84, Regression, Linear; F=0.056
Statistical Analysis 14: Comparison: Parkinson's Disease; Linear Regression of Executive Function Composite Scores and Frontal GE180 SUVR in PD Subjects; Test type: Other — Linear Regression; p = 0.94, Regression, Linear; F=0.008
Statistical Analysis 15: Comparison: Parkinson's Disease; Linear Regression of Speed Composite Scores and Frontal GE180 SUVR in PD Subjects; Test type: Other — Linear Regression; p = 0.29, Regression, Linear; F=2.01
Statistical Analysis 16: Comparison: Parkinson's Disease; Linear Regression of Language Composite Scores and Frontal GE180 SUVR in PD Subjects; Test type: Other — Linear Regression; p = 0.72, Regression, Linear; F=0.173

2. Primary Outcome: Cingulate GE180 Standardized Uptake Value Ratio (SUVR)
Description: Cingulate SUVR- GE180 binding potential in the cingulate ROI, as a marker of cingulate neuroinflammation. Cingulate neuroinflammation would be expected to relate to cingulate AD pathology, and given known cingulate lobe role in executive system function, is hypothesized to relate to measures of executive function in particular, with greater cingulate GE180 relating to poorer cognitive function.
Time Frame: Baseline (Single scan)
Measure: Mean (Standard Deviation); unit: SUVR
Arm/Group | Control | Mild Cognitive Impairment | Alzheimer's Disease | Parkinson's Disease
Number analyzed (Participants) | 10 | 7 | 3 | 4
SUVR | 0.9994 (0.057) | 1.0387 (0.036) | 1.0554 (0.063) | 0.9893 (0.092)
Statistical Analysis 1: Comparison: Control; Linear Regression of Memory Composite Scores and Cingulate GE180 SUVR in Control Subjects; Test type: Other — Linear Regression; p = 0.54, Regression, Linear; F=0.424
Statistical Analysis 2: Comparison: Control; Linear Regression of Executive Function Composite Scores and Cingulate GE180 SUVR in Control Subjects; Test type: Other — Linear Regression; p = 0.53, Regression, Linear; F=0.447
Statistical Analysis 3: Comparison: Control; Linear Regression of Speed Composite Scores and Cingulate GE180 SUVR in Control Subjects; Test type: Other — Linear Regression; p = 0.23, Regression, Linear; F=1.773
Statistical Analysis 4: Comparison: Control; Linear Regression of Language Composite Scores and Cingulate GE180 SUVR in Control Subjects; Test type: Other — Linear Regression; p = 0.01, Regression, Linear; F=3.615
Statistical Analysis 5: Comparison: Mild Cognitive Impairment; Linear Regression of Memory Composite Scores and Cingulate GE180 SUVR in MCI Subjects; Test type: Other — Linear Regression; p = 0.039, Regression, Linear; F=9.204
Statistical Analysis 6: Comparison: Mild Cognitive Impairment; Linear Regression of Executive Function Composite Scores and Cingulate GE180 SUVR in MCI Subjects; Test type: Other — Linear Regression; p = 0.33, Regression, Linear; F=1.209
Statistical Analysis 7: Comparison: Mild Cognitive Impairment; Linear Regression of Speed Composite Scores and Cingulate GE180 SUVR in MCI Subjects; Test type: Other — Linear Regression; p = 0.07, Regression, Linear; F=5.801
Statistical Analysis 8: Comparison: Mild Cognitive Impairment; Linear Regression of Language Composite Scores and Cingulate GE180 SUVR in MCI Subjects; Test type: Other — Linear Regression; p = 0.03, Regression, Linear; F=10.374
Statistical Analysis 9: Comparison: Alzheimer's Disease; Linear Regression of Memory Composite Scores and Cingulate GE180 SUVR in AD Subjects; Test type: Other — Linear Regression; p = 0.27, Regression, Linear; F=5.024
Statistical Analysis 10: Comparison: Alzheimer's Disease; Linear Regression of Executive Function Composite Scores and Cingulate GE180 SUVR in AD Subjects; Test type: Other — Linear Regression; p = 0.16, Regression, Linear; F=15.568
Statistical Analysis 11: Comparison: Alzheimer's Disease; Linear Regression of Speed Composite Scores and Cingulate GE180 SUVR in AD Subjects; Test type: Other — Linear Regression; p = 0.262, Regression, Linear; F=5.238
Statistical Analysis 12: Comparison: Alzheimer's Disease; Linear Regression of Language Composite Scores and Cingulate GE180 SUVR in AD Subjects; Test type: Other — Linear Regression; p = 0.043, Regression, Linear; F=221.308
Statistical Analysis 13: Comparison: Parkinson's Disease; Linear Regression of Memory Composite Scores and Cingulate GE180 SUVR in PD Subjects; Test type: Other — Linear Regression; p = 0.26, Regression, Linear; F=2.430
Statistical Analysis 14: Comparison: Parkinson's Disease; Linear Regression of Executive Function Composite Scores and Cingulate GE180 SUVR in PD Subjects; Test type: Other — Linear Regression; p = 0.38, Regression, Linear; F=1.269
Statistical Analysis 15: Comparison: Parkinson's Disease; Linear Regression of Speed Composite Scores and Cingulate GE180 SUVR in PD Subjects; Test type: Other — Linear Regression; p = 0.07, Regression, Linear; F=13.164
Statistical Analysis 16: Comparison: Parkinson's Disease; Linear Regression of Language Composite Scores and Cingulate GE180 SUVR in PD Subjects; Test type: Other — Linear Regression; p = 0.37, Regression, Linear; F=1.312

3. Primary Outcome: Parietal GE180 Standardized Uptake Value Ratio (SUVR)
Description: Parietal SUVR - GE180 binding potential in the parietal cortical ROI, as a marker of parietal neuroinflammation. Parietal neuroinflammation would be expected to relate to parietal lobe AD pathology, and given known parietal lobe role in visual and executive system function, is hypothesized to relate to measures of visuospatial and executive skills in particular, with greater parietal lobe GE180 relating to poorer cognitive function.
Time Frame: Baseline (Single scan)
Measure: Mean (Standard Deviation); unit: SUVR
Arm/Group | Control | Mild Cognitive Impairment | Alzheimer's Disease | Parkinson's Disease
Number analyzed (Participants) | 10 | 7 | 3 | 4
SUVR | 0.8701 (0.0588) | 0.9241 (0.043) | 0.8847 (0.032) | 0.8562 (0.032)
Statistical Analysis 1: Comparison: Control; Linear Regression of Memory Composite Scores and Parietal GE180 SUVR in Control Subjects; Test type: Other — Linear Regression; p = 0.64, Regression, Linear; F=0.233
Statistical Analysis 2: Comparison: Control; Linear Regression of Executive Function Composite Scores and Parietal GE180 SUVR in Control Subjects; Test type: Other — Linear Regression; p = 0.92, Regression, Linear; F=0.011
Statistical Analysis 3: Comparison: Control; Linear Regression of Speed Composite Scores and Parietal GE180 SUVR in Control Subjects; Test type: Other — Linear Regression; p = 0.22, Regression, Linear; F=1.790
Statistical Analysis 4: Comparison: Control; Linear Regression of Language Composite Scores and Parietal GE180 SUVR in Control Subjects; Test type: Other — Linear Regression; p = 0.42, Regression, Linear; F=0.720
Statistical Analysis 5: Comparison: Mild Cognitive Impairment; Linear Regression of Memory Composite Scores and Parietal GE180 SUVR in MCI Subjects; Test type: Other — Linear Regression; p = 0.61, Regression, Linear; F=0.305
Statistical Analysis 6: Comparison: Mild Cognitive Impairment; Linear Regression of Executive Function Composite Scores and Parietal GE180 SUVR in MCI Subjects; Test type: Other — Linear Regression; p = 0.95, Regression, Linear; F=0.005
Statistical Analysis 7: Comparison: Mild Cognitive Impairment; Linear Regression of Speed Composite Scores and Parietal GE180 SUVR in MCI Subjects; Test type: Other — Linear Regression; p = 0.55, Regression, Linear; F=0.435
Statistical Analysis 8: Comparison: Mild Cognitive Impairment; Linear Regression of Language Composite Scores and Parietal GE180 SUVR in MCI Subjects; Test type: Other — Linear Regression; p = 0.43, Regression, Linear; F=0.787
Statistical Analysis 9: Comparison: Alzheimer's Disease; Linear Regression of Memory Composite Scores and Parietal GE180 SUVR in AD Subjects; Test type: Other — Linear Regression; p = 0.036, Regression, Linear; F=316.379
Statistical Analysis 10: Comparison: Alzheimer's Disease; Linear Regression of Executive Function Composite Scores and Parietal GE180 SUVR in AD Subjects; Test type: Other — Linear Regression; p = 0.39, Regression, Linear; F=2.032
Statistical Analysis 11: Comparison: Alzheimer's Disease; Linear Regression of Speed Composite Scores and Parietal GE180 SUVR in AD Subjects; Test type: Other — Linear Regression; p = 0.031, Regression, Linear; F=425.337
Statistical Analysis 12: Comparison: Alzheimer's Disease; Linear Regression of Language Composite Scores and Parietal GE180 SUVR in AD Subjects; Test type: Other — Linear Regression; p = 0.274, Regression, Linear; F=4.739
Statistical Analysis 13: Comparison: Parkinson's Disease; Linear Regression of Memory Composite Scores and Parietal GE180 SUVR in PD Subjects; Test type: Other — Linear Regression; p = 0.66, Regression, Linear; F=0.263
Statistical Analysis 14: Comparison: Parkinson's Disease; Linear Regression of Executive Function Composite Scores and Parietal GE180 SUVR in PD Subjects; Test type: Other — Linear Regression; p = 0.07, Regression, Linear; F=12.244
Statistical Analysis 15: Comparison: Parkinson's Disease; Linear Regression of Speed Composite Scores and Parietal GE180 SUVR in PD Subjects; Test type: Other — Linear Regression; p = 0.48, Regression, Linear; F=0.762
Statistical Analysis 16: Comparison: Parkinson's Disease; Linear Regression of Language Composite Scores and Parietal GE180 SUVR in PD Subjects; Test type: Other — Linear Regression; p = 0.12, Regression, Linear; F=7.107

4. Primary Outcome: Temporal GE180 Standardized Uptake Value Ratio (SUVR)
Description: Temporal SUVR-- GE180 binding potential in the temporal cortical ROI, as a marker of temporal neuroinflammation. Temporal neuroinflammation would be expected to relate to temporal lobe AD pathology, and given known temporal lobe role in memory and language system function, is hypothesized to relate to measures of memory in particular, with greater temporal lobe GE180 relating to poorer memory and language function.
Time Frame: Baseline (Single scan)
Measure: Mean (Standard Deviation); unit: SUVR
Arm/Group | Control | Mild Cognitive Impairment | Alzheimer's Disease | Parkinson's Disease
Number analyzed (Participants) | 10 | 7 | 3 | 4
SUVR | 0.9127 (0.0668) | 0.9779 (0.046) | 0.9146 (0.045) | 0.8899 (0.056)
Statistical Analysis 1: Comparison: Control; Linear Regression of Memory Composite Scores and Temporal GE180 SUVR in Control Subjects; Test type: Other — Linear Regression; p = 0.85, Regression, Linear; F=0.038
Statistical Analysis 2: Comparison: Control; Linear Regression of Executive Function Composite Scores and Temporal GE180 SUVR in Control Subjects; Test type: Other — Linear Regression; p = 0.84, Regression, Linear; F=0.042
Statistical Analysis 3: Comparison: Control; Linear Regression of Speed Composite Scores and Temporal GE180 SUVR in Control Subjects; Test type: Other — Linear Regression; p = 0.35, Regression, Linear; F=1.021
Statistical Analysis 4: Comparison: Control; Linear Regression of Language Composite Scores and Temporal GE180 SUVR in Control Subjects; Test type: Other — Linear Regression; p = 0.25, Regression, Linear; F=1.610
Statistical Analysis 5: Comparison: Mild Cognitive Impairment; Linear Regression of Memory Composite Scores and Temporal GE180 SUVR in MCI Subjects; Test type: Other — Linear Regression; p = 0.25, Regression, Linear; F=1.779
Statistical Analysis 6: Comparison: Mild Cognitive Impairment; Linear Regression of Executive Function Composite Scores and Temporal GE180 SUVR in MCI Subjects; Test type: Other — Linear Regression; p = 0.54, Regression, Linear; F=0.455
Statistical Analysis 7: Comparison: Mild Cognitive Impairment; Linear Regression of Speed Composite Scores and Temporal GE180 SUVR in MCI Subjects; Test type: Other — Linear Regression; p = 0.47, Regression, Linear; F=0.650
Statistical Analysis 8: Comparison: Mild Cognitive Impairment; Linear Regression of Language Composite Scores and Temporal GE180 SUVR in MCI Subjects; Test type: Other — Linear Regression; p = 0.74, Regression, Linear; F=0.131
Statistical Analysis 9: Comparison: Alzheimer's Disease; Linear Regression of Memory Composite Scores and Temporal GE180 SUVR in AD Subjects; Test type: Other — Linear Regression; p = 0.83, Regression, Linear; F=0.075
Statistical Analysis 10: Comparison: Alzheimer's Disease; Linear Regression of Executive Function Composite Scores and Temporal GE180 SUVR in AD Subjects; Test type: Other — Linear Regression; p = 0.41, Regression, Linear; F=1.831
Statistical Analysis 11: Comparison: Alzheimer's Disease; Linear Regression of Speed Composite Scores and Temporal GE180 SUVR in AD Subjects; Test type: Other — Linear Regression; p = 0.83, Regression, Linear; F=0.079
Statistical Analysis 12: Comparison: Alzheimer's Disease; Linear Regression of Language Composite Scores and Temporal GE180 SUVR in AD Subjects; Test type: Other — Linear Regression; p = 0.52, Regression, Linear; F=0.879
Statistical Analysis 13: Comparison: Parkinson's Disease; Linear Regression of Memory Composite Scores and Temporal GE180 SUVR in PD Subjects; Test type: Other — Linear Regression; p = 0.98, Regression, Linear; F=0.001
Statistical Analysis 14: Comparison: Parkinson's Disease; Linear Regression of Executive Function Composite Scores and Temporal GE180 SUVR in PD Subjects; Test type: Other — Linear Regression; p = 0.95, Regression, Linear; F=0.005
Statistical Analysis 15: Comparison: Parkinson's Disease; Linear Regression of Speed Composite Scores and Temporal GE180 SUVR in PD Subjects; Test type: Other — Linear Regression; p = 0.32, Regression, Linear; F=1.733
Statistical Analysis 16: Comparison: Parkinson's Disease; Linear Regression of Language Composite Scores and Temporal GE180 SUVR in PD Subjects; Test type: Other — Linear Regression; p = 0.67, Regression, Linear; F=0.249

5. Primary Outcome: Whole Brain GE180 Standardized Uptake Value Ratio (SUVR)
Description: Whole Brain GE180- GE180 binding potential in the whole brain, as a marker of global neuroinflammation. Global neuroinflammation would be expected to relate to more widespread pathology on average, and is hypothesized to relate to global measures of cognition, including the MoCA and DRS, with greater whole brain GE180 relating to poorer cognitive function overall.
Time Frame: Baseline (Single scan)
Measure: Mean (Standard Deviation); unit: SUVR
Arm/Group | Control | Mild Cognitive Impairment | Alzheimer's Disease | Parkinson's Disease
Number analyzed (Participants) | 10 | 7 | 3 | 4
SUVR | 0.9179 (0.0545) | 0.9711 (0.034) | 0.9351 (0.010) | 0.9051 (0.046)
Statistical Analysis 1: Comparison: Control; Linear Regression of DRS Scores and Whole Brain GE180 SUVR in Control Subjects; Test type: Other — Linear Regression; p = 0.76, Regression, Linear; F=0.098
Statistical Analysis 2: Comparison: Control; Linear Regression of MoCA Scores and Whole Brain GE180 SUVR in Control Subjects; Test type: Other — Linear Regression; p = 0.49, Regression, Linear; F=0.513
Statistical Analysis 3: Comparison: Mild Cognitive Impairment; Linear Regression of DRS Scores and Whole Brain GE180 SUVR in MCI Subjects; Test type: Other — Linear Regression; p = 0.93, Regression, Linear; F=0.008
Statistical Analysis 4: Comparison: Mild Cognitive Impairment; Linear Regression of MoCA Scores and Whole Brain GE180 SUVR in MCI Subjects; Test type: Other — Linear Regression; p = 0.54, Regression, Linear; F=0.430
Statistical Analysis 5: Comparison: Alzheimer's Disease; Linear Regression of DRS Scores and Whole Brain GE180 SUVR in AD Subjects; Test type: Other — Linear Regression; p = 0.77, Regression, Linear; F=0.142
Statistical Analysis 6: Comparison: Alzheimer's Disease; Linear Regression of MoCA Scores and Whole Brain GE180 SUVR in AD Subjects; Test type: Other — Linear Regression; p = 0.61, Regression, Linear; F=0.496
Statistical Analysis 7: Comparison: Parkinson's Disease; Linear Regression of DRS Scores and Whole Brain GE180 SUVR in PD Subjects; Test type: Other — Linear Regression; p = 0.11, Regression, Linear; F=8.046
Statistical Analysis 8: Comparison: Parkinson's Disease; Linear Regression of MoCA Scores and Whole Brain GE180 SUVR in PD Subjects; Test type: Other — Linear Regression; p = 0.84, Regression, Linear; F=0.051

6. Primary Outcome: Memory Composite Score (Z-score)
Description: The memory composite score is comprised from data from two gold-standard clinical measures of verbal and nonverbal memory (Rey Auditory Verbal Learning Test, delayed recall score; Brief Visuospatial Memory Test, Revised, delayed recall score). The raw score for each individual assessment is corrected for age based on published normative data for each test. These adjusted scores (T scores and/or scaled scores) are converted to z-scores, then the two z-scores are averaged together to create the composite score. A higher value is indicative of better memory function, a lower value is indicative of worse memory function. A z-score of 0 represents the sample mean. Composite Z-scores do not have direct clinical relevance.
Time Frame: Baseline (Pre-scan)
Measure: Mean (Standard Deviation); unit: z score
Arm/Group | Control | Mild Cognitive Impairment | Alzheimer's Disease | Parkinson's Disease
Number analyzed (Participants) | 10 | 7 | 3 | 4
z score | 0.367 (0.86) | -0.675 (1.42) | -2.483 (0.35) | -0.404 (0.88)

7. Primary Outcome: Executive Function Composite Score (Z-score)
Description: The executive function composite score is comprised from data from two gold-standard clinical measures of set-shifting and inhibition (Trail Making Test, part B; Delis Kaplan Executive Functioning Scale Color Word Inhibition, inhibition score). The raw score for each individual assessment is corrected for age based on published normative data for each test. These adjusted scores (T scores and/or scaled scores) are converted to z-scores, then the two z-scores are averaged together to create the composite score. A higher value is indicative of better executive function, a lower value is indicative of worse executive function. A z-score of 0 represents the sample mean. Composite Z-scores do not have direct clinical relevance.
Time Frame: Baseline (Pre-scan)
Measure: Mean (Standard Deviation); unit: z score
Arm/Group | Control | Mild Cognitive Impairment | Alzheimer's Disease | Parkinson's Disease
Number analyzed (Participants) | 10 | 7 | 3 | 4
z score | 0.572 (0.90) | -0.011 (0.42) | -1.361 (1.99) | 0.029 (0.90)

8. Primary Outcome: Speed Composite Score (Z-score)
Description: The speed composite score is comprised from data from two gold-standard clinical measures of speeded attention and psychomotor speed (Trail Making Test, part A; Symbol Digit Modalities Test, oral version). The raw score for the Symbol Digit Modalities Test, oral version is converted directly to a z-score based on published normative data. The Trail making Test, part A is corrected for age based on published normative data, resulting in a T-score, which is then converted to a z-score. Then the two z-scores are averaged together to create the composite score. A higher value is indicative of better speed function, a lower value is indicative of worse speed function. A z-score of 0 represents the sample mean. Composite Z-scores do not have direct clinical relevance.
Time Frame: Baseline (Pre-scan)
Measure: Mean (Standard Deviation); unit: z score
Arm/Group | Control | Mild Cognitive Impairment | Alzheimer's Disease | Parkinson's Disease
Number analyzed (Participants) | 10 | 7 | 3 | 4
z score | 0.285 (1.28) | -0.013 (0.78) | -1.585 (1.06) | -0.731 (0.60)

9. Primary Outcome: Language Composite Score (Z-score)
Description: The language composite score is comprised from data from two gold-standard clinical measures of confrontation naming and semantic fluency (Boston Naming Test; Animal Naming Test). The raw score for the Animal Naming Test is converted directly to a z-score based on published normative data. The Boston Naming Test is corrected for age based on published normative data, resulting in a scaled score, which is then converted to a z-score. Then the two z-scores are averaged together to create the composite score. A higher value is indicative of better language function, a lower value is indicative of worse language function. A z-score of 0 represents the sample mean. Composite Z-scores do not have direct clinical relevance.
Time Frame: Baseline (Pre-scan)
Measure: Mean (Standard Deviation); unit: z score
Arm/Group | Control | Mild Cognitive Impairment | Alzheimer's Disease | Parkinson's Disease
Number analyzed (Participants) | 10 | 7 | 3 | 4
z score | 0.584 (0.857) | -0.234 (1.12) | -0.7272 (0.92) | 0.541 (1.18)

10. Primary Outcome: Dementia Rating Score
Description: DRS- The Dementia Rating Scale is a comprehensive, but relatively brief assessment of overall cognitive functioning. The measure consists of items testing memory, attention, executive skills, and visuospatial skill, for a total of 144 points. A score of less than 124 is indicative of dementia level cognitive functioning. A higher score indicates a better outcome.
Time Frame: Baseline (Pre-scan)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Mild Cognitive Impairment | Alzheimer's Disease | Parkinson's Disease
Number analyzed (Participants) | 10 | 7 | 3 | 4
score on a scale | 139.2 (2.97) | 130.4 (3.87) | 120.3 (12.42) | 139.3 (5.25)

11. Primary Outcome: Montreal Cognitive Assessment Score (MoCA)
Description: MoCA -The Montreal Cognitive Assessment is a brief screening tool, originally designed to detect patients with MCI in a memory disorders clinic [10]. Standard administration consists of 12 individual tasks grouped into seven cognitive domains (visuospatial/executive, naming; attention, language, abstraction, memory, and orientation). Task performance is summed generating both domain and a total score. An education correction of one point is added to the total score for individuals with 12 years of education or less. Scores range from 0-30, with a score of 26 or less indicating cognitive impairment.
Time Frame: Baseline (Pre-scan)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Mild Cognitive Impairment | Alzheimer's Disease | Parkinson's Disease
Number analyzed (Participants) | 10 | 7 | 3 | 4
score on a scale | 26.0 (2.36) | 23.4 (2.44) | 18.3 (4.73) | 27.5 (1.00)

ADVERSE EVENTS:
Time Frame: 24 hours
Description: There was no anticipated risk of mortality (all-causes) during the course of the project.
Arm/Group | Control | Mild Cognitive Impairment | Alzheimer's Disease | Parkinson's Disease
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/7 | 0/3 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/7 | 0/3 | 0/4
Other Adverse Events (participants affected / at risk) | 1/10 | 2/7 | 1/3 | 0/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=10) | Mild Cognitive Impairment (N=7) | Alzheimer's Disease (N=3) | Parkinson's Disease (N=4)
Low-Grade Headache (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Mild Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Limitations of the data presented here include reduced power in the statistical analysis due to reduced enrollment, and should be reviewed in the context of recent data related to the blood-brain barrier permeability of GE180.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-03): https://cdn.clinicaltrials.gov/large-docs/16/NCT03702816/Prot_SAP_000.pdf